CLINICAL TRIAL: NCT06688903
Title: EMPOWERing Patients With Chronic Diseases Through Smartphone App, Health Coaching and Community-based Intervention
Brief Title: App-based Diabetes Management and Community-based Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202409-00001
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: App-based diabetes management and community-based health coaching

INTERVENTIONS:
Behavioral: App-based diabetes management and community-based health coaching — All participants will use the EMPOWER+ app and a Fitbit wearable. They will also received community-based health coaching and/or other prescribed structured programmes.

SUMMARY:
Community-based health coaching interventions play a vital role in complementing the traditional chronic disease management model for type 2 diabetes patients. Compared to conventional approaches that often focus on periodic clinical visits, community-based coaching could provide continuous, personalised support within patients in everyday environments. Health coaches work directly with patients to set realistic goals, develop individualised action plans, and provide ongoing motivation and accountability. This personalised attention helps to improve self-management skills, such as medication adherence, dietary choices, and physical activity, which are crucial for chronic disease management and preventing complications. Our mobile health app, EMPOWER+ has multiple logging features, gamified elements to help users set goals and provide rewards, educational resources, and personalised nudges generated based on real users; inputs and predictive modeling. It has demonstrated some preliminary effectiveness and acceptability within the clinical settings. This trial aims to assess its effectiveness, adoption, and sustainability in the less-controlled community settings, preparing for its large implementation in the future.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years and above
* Having been diagnosed with type 2 diabetes mellitus
* Having most recent HbA1c ≥ 6.5%
* Physically able to exercise
* Able to read, write, and converse in English
* Able to comply with study procedures

Exclusion Criteria:

* Requiring assistance with basic activities of daily living (BADL)
* Have planned major operation or surgical procedure within 6 months from the time of recruitment
* Current pregnant or lactating

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months
  HbA1c over 6 months

SECONDARY OUTCOMES:
Physical activity as measured by number of steps | 6 months
  Physical activity over 6 months
Physical activity as measured by moderate to vigorous active minutes | 6 months
  Physical activity over 6 months
Physical activity as measured by GPAQ | 6 months
  Physical activity as measured by GPAQ
Patient activation score as measured by patient activation measure | 6 months
  Difference in patient activation score between intervention and control over 6 months
Medication adherence as measured by MARS-5 | 6 months
  Difference in medication adherence between intervention and control over 6 months
Quality of life as measured by EQ-5D-5L | 6 months
  Difference in quality of life between intervention and control over 6 months
Healthcare cost as measured by cost of consultations, lab tests, medications, admission | 6 months
  Healthcare cost over 6 months
Healthcare cost as measured by WPAI | 6 months
  Healthcare cost over 6 months
Maintenance of the intervention effects on HbA1c | 6 months
  HbA1c over 6 months after the 6-month intervention
Maintenance of the intervention effects on blood pressure | 6 months
  Blood pressure over 6 months after the 6-month intervention
Maintenance of the intervention effects on total cholesterol | 6 months
  Total cholesterol over 6 months after the 6-month intervention
Maintenance of the intervention effects on high-density lipoprotein (HDL) | 6 months
  HDL over 6 months after the 6-month intervention
Maintenance of the intervention effects on low-density lipoprotein (LDL) | 6 months
  LDL over 6 months after the 6-month intervention
Maintenance of the intervention effects on triglycerides | 6 months
  Triglycerides over 6 months after the 6-month intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore